CLINICAL TRIAL: NCT06256354
Title: Effects of Intraoperative Targeted Temperature Management on Incidence of Postoperative Delirium and Long-term Survival in Older Patients Having Major Cancer Surgery: A Multicenter Randomized Trial
Brief Title: Effects of Intraoperative Targeted Temperature Management on Incidence of Postoperative Delirium and Long-term Survival
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-185
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cancer Surgery; Hypothermia; Delirium; Long-term Survivors
Keywords: Cancer surgery; Hypothermia; Delirium; Long-term survival
MeSH Terms: conditions — Hypothermia; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine thermal management (Placebo Comparator): Patients assigned to routine thermal management will not be pre-warmed and ambient intraoperative temperature will be maintained near 20°C per routine. Only transfused blood will be warmed. An upper- or lower-body forced-air cover will be positioned over an appropriate non-operative site but will not initially be activated. Should core temperature decrease to 35.5°C, the warmer will be activated as necessary to prevent core temperature from decreasing further. The target nasopharyngeal temperature is 35.5°C.
  Interventions: Other: Routine thermal management
- Target temperature management (Experimental): Pre-warming is performed with a full-body forced-air cover and electrically heated blanket for about 30 minutes before induction of anesthesia. The warmer will initially be set to "high" which corresponds to about 43°C. It will be subsequently adjusted to make patients feel warm, but not uncomfortably so. Patients will be warmed during surgery using two forced-air covers or combining forced-air covers with electric heating blanket when clinically practical. All intravenous fluids will be warmed to body temperature. There is no need to control ambient temperature since ambient temperature has little effect on core temperature in patients warmed with forced air. The target nasopharyngeal temperature is 36.8°C.
  Interventions: Other: Target temperature management

INTERVENTIONS:
Other: Routine thermal management — Patients assigned to routine thermal management will not be pre-warmed and ambient intraoperative temperature will be maintained near 20°C per routine. Only transfused blood will be warmed. An upper- or lower-body forced-air cover will be positioned over an appropriate non-operative site but will not initially be activated. Should core temperature decrease to 35.5°C, the warmer will be activated as necessary to prevent core temperature from decreasing further. The target nasopharyngeal temperature is 35.5°C.
  Arms: Routine thermal management
Other: Target temperature management — Pre-warming is performed with a full-body forced-air cover and electrically heated blanket for about 30 minutes before induction of anesthesia. The warmer will initially be set to "high" which corresponds to about 43°C. It will be subsequently adjusted to make patients feel warm, but not uncomfortably so. Patients will be warmed during surgery using two forced-air covers or combining forced-air covers with electric heating blanket when clinically practical. All intravenous fluids will be warmed to body temperature. There is no need to control ambient temperature since ambient temperature has little effect on core temperature in patients warmed with forced air. The target nasopharyngeal temperature is 36.8℃.
  Arms: Target temperature management

SUMMARY:
Intraoperative hypothermia is common in patients having major surgery and the compliance with intraoperative temperature monitoring and management remains poor. Studies suggest that intraoperative hypothermia is an important risk factor of postoperative delirium, which is associated with worse early and long-term outcomes. Furthermore, perioperative hypothermia increases stress responses and provokes immune suppression, which might promote cancer recurrence and metastasis. In a recent trial, targeted temperature management reduced intraoperative hypothermia and emergence delirium. There was also a trend of reduced postoperative delirium, although not statistically significant. This trial is designed to test the hypothesis that intraoperative targeted temperature management may reduce postoperative delirium and improves progression-free survival in older patients recovering from major cancer surgery.

DETAILED DESCRIPTION:
Perioperative hypothermia results from anesthetic-impaired thermoregulatory responses combined with cool operating rooms and exposed body cavities. Core temperatures <35.5°C increases perioperative blood loss, delays post anesthetic recovery, and increases surgical wound infections.

Despite guideline recommendations, compliance with intraoperative temperature monitoring and management remains poor. In a national survey published in 2017, intraoperative hypothermia (core temperature <36.0°C) occurred in 44% of patients having elective surgery with general anesthesia. According to a survey of anesthesiologists in six Asia-Pacific countries (Singapore, Malaysia, Philippines, Thailand, India, and South Korea), only 67% of respondents measured temperature intraoperatively during general anesthesia, and only 44% report intraoperative active warming and warming was ineffective in more than half of their patients. Perioperative hypothermia thus remains common.

The 5,056-patient PROTECT trial showed that myocardial injury, surgical site infections, and blood loss were similar in patients randomized to intraoperative core temperatures of 35.5 or 37°C. However, there are other important complications that may be caused by intraoperative hypothermia including delirium, cancer recurrence, shivering, and thermal discomfort.

Perioperative neurocognitive disorders (NCDs), especially postoperative delirium and postoperative cognitive dysfunction (POCD), are significant challenges to older patients scheduled for surgery. Delirium is a syndrome of acutely occurring and fluctuating changes in attention, level of consciousness, and cognitive function. Postoperative cognitive dysfunction refers to cognitive decline (including the ability of study, memory, action, and judgement) detected from 30 days to 12 months after surgery.

In patients aged 60 years or above, the incidence of postoperative delirium is about 12-24%. The incidence of POCD is about 7-12% at 3-month follow-up and is associated with delirium, although the relationship is probably not causal. Delirium and POCD are associated with worse perioperative outcomes including prolonged hospitalization, increased complications, and high mortality, and worse long-term outcomes including shortened overall survival, as well as increased dementia and lowered life quality.

Postoperative delirium and POCD are multifactorial. Predisposing factors include advanced age, lower educational level, cognitive impairment, comorbidities (e.g., cerebrovascular disease, diabetes, and kidney disease), alcohol abuse, and malnutrition. Precipitating factors include deep anesthesia, opioid use, benzodiazepines, intraoperative blood loss/blood transfusion, and severe pain. Hypothermia may also increase the risk of delirium.

Hypothermia provokes both autonomic and behavioral protective responses. The first autonomic response is arterio-venous shunt constriction. Thermoregulatory vasoconstriction occurs many times a day in a typical hospital environment. It is highly effective, but does not usually disturb people and is generally considered to be of little consequence. Shivering is the other primary autonomic thermoregulatory defense against cold and has a triggering threshold about 1°C below the core temperature that triggers vasoconstriction. Unlike vasoconstriction, shivering is uncomfortable for patients. Furthermore, it is accompanied by a tripling of catecholamine concentrations, hypertension, and tachycardia. Behavioral thermoregulatory defenses are mediated by thermal comfort, and provoke voluntary defensive measures such as putting on a sweater, open windows, etc. Behavioral defenses include air conditioning and building shelters and are thus far stronger than autonomic responses. Thermal comfort matters to patients and is thus worth evaluating.

Despite advances in surgery and oncology, postoperative survival decreases about 10% per year, mainly due to cancer recurrence. The development of cancer recurrence mainly depends on the balance between the invasive ability of residual cancer cells and the anti-cancer immune function. Perioperative hypothermia increases stress responses and provokes immune suppression.

The investigators therefore propose to determine whether intraoperative targeted temperature management decreases the incidence of delirium, improves thermal comfort, reduces postoperative shivering, and improves long-term survival in older patients recovering from major cancer surgery. Specifically, the investigators will test the primary short-term hypothesis that perioperative normothermia (core temperature near 36.8°C) reduces delirium over the initial 4 postoperative days. Secondary short-term hypotheses are that perioperative normothermia improves thermal comfort, reduces shivering, reduces incidence of emergence delirium, and reduces blood transfusion. The primary long-term hypothesis is that perioperative normothermia improves progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years.
2. Planned potentially curative initial cancer surgery with an expected duration of 2 hours or longer under general anesthesia.

Exclusion Criteria:

1. Preoperative fever (tympanic temperature ≥38℃).
2. Known or suspected preoperative infection.
3. Previous history of schizophrenia, epilepsy, Parkinson disease, myasthenia gravis, or delirium.
4. Unable to communicate due to severe dementia, language barrier, or coma.
5. Critically ill (Left ventricular ejection fraction <30%, Child-Pugh grades C, requirement of renal replacement therapy, American Society of Anesthesiologists physical status>IV, or expected survival <24 hours).
6. Scheduled surgery for breast cancer, intracranial tumors, or rare cancers.
7. Planned to undergo therapeutic hypothermia.
8. Body mass index >30 kg/m2 (to facilitate thermal management).
9. Have participated in this study previously.
10. Any other conditions that are considered unsuitable for study participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3992 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within 4 days after surgery | During the first four days after surgery.
  Occurrence of delirium during the first four postoperative days is assessed with the 3D-Confusion Assessment Method (3D-CAM) or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU; for intubated patients) twice daily (8-10 am and 6-8 pm). Any positive CAM evaluation will be considered evidence of delirium. Immediately before assessing delirium, sedation or agitation is assessed with the Richmond Agitation-Sedation Scale (RASS; scores range from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm). Deeply sedated or unarousable patients (RASS -4 or -5) is recorded as comatose and not assessed for delirium.
Progression-free survival after surgery [long-term] | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer recurrence/metastasis/progression or all-cause death, whichever comes first.

SECONDARY OUTCOMES:
Postoperative thermal comfort | Up to 30 minutes after arriving PACU/ICU or after extubation.
  Postoperative thermal comfort is evaluated with the Numerical Rating Scale (NRS; an 11-point scale where 0=intense cold, 5=thermal comfort, and 10=intense warm). For patients who are extubated in the operation room, evaluation is conducted at 5 and 30 minutes after arriving post-anesthesia care unit (PACU)/intensive care unit (ICU). For patients who are admitted to PACU/ICU with endotracheal intubation, evaluation is conducted at 5 and 30 minutes after extubation. If patients remain intubated 2 hours after surgery, no further thermal comfort assessments will be conducted.
Postoperative shivering intensity | Up to 30 minutes after arriving PACU/ICU or after extubation.
  Postoperative shivering intensity is evaluated with a four-point scale (0=no shivering, 1=intermittent, mild shivering, 2=moderate shivering, and 3=persistent, intense shivering). For patients who are extubated in the operation room, evaluation is conducted at 5 and 30 minutes after arriving post-anesthesia care unit (PACU)/intensive care unit (ICU). For patients who are admitted to PACU/ICU with endotracheal intubation, evaluation is conducted at 5 and 30 minutes after extubation. If patients remain intubated 2 hours after surgery, no further shivering assessments will be conducted.
Incidence of emergence delirium | Up to 30 minutes after arriving PACU/ICU or after extubation.
  Patients are firstly be evaluated with the Richmond Agitation-Sedation Scale (RASS; scores range from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm). Patients will then be evaluated with the Confusion Assessment Method (CAM-ICU) for the Intensive Care Unit. For patients who are extubated in the operation room, evaluation is conducted at 5 and 30 minutes after arriving post-anesthesia care unit (PACU)/intensive care unit (ICU). For patients who are admitted to PACU/ICU with endotracheal intubation, evaluation is conducted at 5 and 30 minutes after extubation. If patients remain intubated 2 hours after surgery, no further emergence delirium assessments will be conducted.
Units of blood transfused during and within 4 days of surgery | Up to 4 days after surgery.
  Units of blood transfused during surgery and the first 4 days after surgery.
Incidence of postoperative neurocognitive disorders at 6 months after surgery [long-term] | At 6 months after surgery.
  Cognitive function will be assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) before surgery and at 6 months after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline will be considered as the occurrence of postoperative neurocognitive disorders.
Cancer-specific survival after surgery [long-term] | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer-specific death, with deaths from other causes being censored at the time of death. Cancer-specific death is defined as death fully attributable to the cancer for which the index surgery is performed and usually involves cancer recurrence/metastasis/progression after exclusion of other causes such as stroke and myocardial infarction.

OTHER OUTCOMES:
Length of stay in post-anesthesia care unit (PACU) | Up to 24 hours after surgery.
  Length of stay in post-anesthesia care unit (PACU)
Quality of Recovery-15 score on the first day after surgery | Up to 24 hours after surgery.
  Quality of recovery is assessed with the Quality of Recovery-15 questionaire in the first postoperative day.
Change in hemoglobin from baseline (last preoperative concentration) to the lowest concentration on the first day after surgery | Up to 24 hours after surgery.
  Change in hemoglobin from baseline (last preoperative concentration) to the lowest concentration on the first day after surgery
Postoperative duration of hospitalization | Up to 30 days after surgery.
  Postoperative duration of hospitalization
Incidence of delayed neurocognitive recovery on the 30th day after surgery. | At 30 days after surgery.
  Cognitive function will be assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) before surgery and at 30 days after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline will be considered the occurrence of delayed neurocognitive recovery.
Incidence of superficial and serious surgical site infections with 30 days after surgery. | Up to 30 days after surgery.
  Serious infections will include deep and organ-space infections, anastomotic leaks, wound dehiscence, abscess, and sepsis. The definitions were modified from "Guideline for prevention of surgical site infection, 1999" (https://stacks.cdc.gov/view/cdc/7160).
Incidence of non-delirium major complications within 30 days after surgery. | Up to 30 days after surgery
  Non-delirium major complications are defined as new-onset medical events other than delirium that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
All-cause 30-day mortality | Up to 30 days after surgery.
  All-cause 30-day mortality
Incidence of postoperative neurocognitive disorders at 1 year after surgery [long-term] | At 1 year after surgery.
  Cognitive function will be assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) before surgery and at 1 year after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline will be considered as the occurrence of postoperative neurocognitive disorders.
Overall survival after surgery [long-term] | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to all-cause death.
Event-free survival after surgery [long-term] | Up to 3 years after surgery of the last enrolled patient.
  Time interval from index surgery to cancer recurrence/metastasis/progression, new-onset cancer, new-onset serious illness (requiring hospitalization), or all-cause death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (34):
- China (34):
  - The People's Hospital of Chizhou, Chizhou, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Maanshan People's Hospital, Ma’anshan, Anhui
  - Dongzhimen Hospital Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Aerospace Medical Center, Beijing, Beijing Municipality
  - Beijing Chuanyangliu Hospital, Beijing, Beijing Municipality
  - Beijing Coal Group General Hospital, Beijing, Beijing Municipality
  - Beijing Electric Power Hospital, Beijing, Beijing Municipality
  - The First Hospital of Tsinghua University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Fourth Hospital of Hebei Medical University (Hebei Tumor Hospital), Shijiazhuang, Hebei
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - The First Affiliated Hospital of Kangda College of Nanjing Medical University ( Lianyungang First People's Hospital), Lianyungang, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The People's Hospital of Wuxi, Wuxi, Jiangsu
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital Of Shandong First Medical University, Jinan, Shandong
  - The People's Hospital of Liaocheng, Liaocheng, Shandong
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - The Second People's Hospital of Yibin (affiliated with West China Hospital of Sichuan University), Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horosz B, Adamiec A, Malec-Milewska M, Misiolek H. Guidelines of the Polish Society of Anaesthesiology and Intensive Therapy regarding prevention of inadvertent intraoperative hypothermia. Anaesthesiol Intensive Ther. 2021;53(5):376-385. doi: 10.5114/ait.2021.111871. PMID 35100795
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Reynolds L, Beckmann J, Kurz A. Perioperative complications of hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):645-57. doi: 10.1016/j.bpa.2008.07.005. PMID 19137808
- [Background] Yi J, Lei Y, Xu S, Si Y, Li S, Xia Z, Shi Y, Gu X, Yu J, Xu G, Gu E, Yu Y, Chen Y, Jia H, Wang Y, Wang X, Chai X, Jin X, Chen J, Xu M, Xiong J, Wang G, Lu K, Yu W, Lei W, Qin Z, Xiang J, Li L, Xiang Z, Pan S, Zhan L, Qiu K, Yao M, Huang Y. Intraoperative hypothermia and its clinical outcomes in patients undergoing general anesthesia: National study in China. PLoS One. 2017 Jun 8;12(6):e0177221. doi: 10.1371/journal.pone.0177221. eCollection 2017. PMID 28594825
- [Background] Koh W, Chakravarthy M, Simon E, Rasiah R, Charuluxananan S, Kim TY, Chew STH, Brauer A, Ti LK. Perioperative temperature management: a survey of 6 Asia-Pacific countries. BMC Anesthesiol. 2021 Aug 16;21(1):205. doi: 10.1186/s12871-021-01414-6. PMID 34399681
- [Background] Sun Z, Honar H, Sessler DI, Dalton JE, Yang D, Panjasawatwong K, Deroee AF, Salmasi V, Saager L, Kurz A. Intraoperative core temperature patterns, transfusion requirement, and hospital duration in patients warmed with forced air. Anesthesiology. 2015 Feb;122(2):276-85. doi: 10.1097/ALN.0000000000000551. PMID 25603202
- [Background] Sessler DI, Pei L, Li K, Cui S, Chan MTV, Huang Y, Wu J, He X, Bajracharya GR, Rivas E, Lam CKM; PROTECT Investigators. Aggressive intraoperative warming versus routine thermal management during non-cardiac surgery (PROTECT): a multicentre, parallel group, superiority trial. Lancet. 2022 May 7;399(10337):1799-1808. doi: 10.1016/S0140-6736(22)00560-8. Epub 2022 Apr 4. PMID 35390321
- [Background] Kong H, Xu LM, Wang DX. Perioperative neurocognitive disorders: A narrative review focusing on diagnosis, prevention, and treatment. CNS Neurosci Ther. 2022 Aug;28(8):1147-1167. doi: 10.1111/cns.13873. Epub 2022 Jun 1. PMID 35652170
- [Background] Silva AR, Regueira P, Albuquerque E, Baldeiras I, Cardoso AL, Santana I, Cerejeira J. Estimates of Geriatric Delirium Frequency in Noncardiac Surgeries and Its Evaluation Across the Years: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2021 Mar;22(3):613-620.e9. doi: 10.1016/j.jamda.2020.08.017. Epub 2020 Oct 1. PMID 33011097
- [Background] Berian JR, Zhou L, Russell MM, Hornor MA, Cohen ME, Finlayson E, Ko CY, Rosenthal RA, Robinson TN. Postoperative Delirium as a Target for Surgical Quality Improvement. Ann Surg. 2018 Jul;268(1):93-99. doi: 10.1097/SLA.0000000000002436. PMID 28742701
- [Background] Goldberg TE, Chen C, Wang Y, Jung E, Swanson A, Ing C, Garcia PS, Whittington RA, Moitra V. Association of Delirium With Long-term Cognitive Decline: A Meta-analysis. JAMA Neurol. 2020 Nov 1;77(11):1373-1381. doi: 10.1001/jamaneurol.2020.2273. PMID 32658246
- [Background] Huang H, Li H, Zhang X, Shi G, Xu M, Ru X, Chen Y, Patel MB, Ely EW, Lin S, Zhang G, Zhou J. Association of postoperative delirium with cognitive outcomes: A meta-analysis. J Clin Anesth. 2021 Dec;75:110496. doi: 10.1016/j.jclinane.2021.110496. Epub 2021 Sep 2. PMID 34482263
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Gleason LJ, Schmitt EM, Kosar CM, Tabloski P, Saczynski JS, Robinson T, Cooper Z, Rogers SO Jr, Jones RN, Marcantonio ER, Inouye SK. Effect of Delirium and Other Major Complications on Outcomes After Elective Surgery in Older Adults. JAMA Surg. 2015 Dec;150(12):1134-40. doi: 10.1001/jamasurg.2015.2606. PMID 26352694
- [Background] Crocker E, Beggs T, Hassan A, Denault A, Lamarche Y, Bagshaw S, Elmi-Sarabi M, Hiebert B, Macdonald K, Giles-Smith L, Tangri N, Arora RC. Long-Term Effects of Postoperative Delirium in Patients Undergoing Cardiac Operation: A Systematic Review. Ann Thorac Surg. 2016 Oct;102(4):1391-9. doi: 10.1016/j.athoracsur.2016.04.071. Epub 2016 Jun 22. PMID 27344279
- [Background] Pereira JV, Aung Thein MZ, Nitchingham A, Caplan GA. Delirium in older adults is associated with development of new dementia: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2021 Jul;36(7):993-1003. doi: 10.1002/gps.5508. Epub 2021 Feb 27. PMID 33638566
- [Background] Zhang Y, He ST, Nie B, Li XY, Wang DX. Emergence delirium is associated with increased postoperative delirium in elderly: a prospective observational study. J Anesth. 2020 Oct;34(5):675-687. doi: 10.1007/s00540-020-02805-8. Epub 2020 Jun 7. PMID 32507939
- [Background] Wagner D, Hooper V, Bankieris K, Johnson A. The Relationship of Postoperative Delirium and Unplanned Perioperative Hypothermia in Surgical Patients. J Perianesth Nurs. 2021 Feb;36(1):41-46. doi: 10.1016/j.jopan.2020.06.015. Epub 2020 Oct 14. PMID 33067117
- [Background] Xu G, Li T, Huang Y. The Effects of Intraoperative Hypothermia on Postoperative Cognitive Function in the Rat Hippocampus and Its Possible Mechanisms. Brain Sci. 2022 Jan 12;12(1):96. doi: 10.3390/brainsci12010096. PMID 35053838
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Lopez M, Sessler DI, Walter K, Emerick T, Ozaki M. Rate and gender dependence of the sweating, vasoconstriction, and shivering thresholds in humans. Anesthesiology. 1994 Apr;80(4):780-8. doi: 10.1097/00000542-199404000-00009. PMID 8024131
- [Background] Kurz A, Sessler DI, Birnbauer F, Illievich UM, Spiss CK. Thermoregulatory vasoconstriction impairs active core cooling. Anesthesiology. 1995 Apr;82(4):870-6. doi: 10.1097/00000542-199504000-00008. PMID 7717557
- [Background] Kurz A, Sessler DI, Christensen R, Dechert M. Heat balance and distribution during the core-temperature plateau in anesthetized humans. Anesthesiology. 1995 Sep;83(3):491-9. doi: 10.1097/00000542-199509000-00007. PMID 7661349
- [Background] Kurz A, Go JC, Sessler DI, Kaer K, Larson MD, Bjorksten AR. Alfentanil slightly increases the sweating threshold and markedly reduces the vasoconstriction and shivering thresholds. Anesthesiology. 1995 Aug;83(2):293-9. doi: 10.1097/00000542-199508000-00009. PMID 7631951
- [Background] Kurz A, Sessler DI, Narzt E, Bekar A, Lenhardt R, Huemer G, Lackner F. Postoperative hemodynamic and thermoregulatory consequences of intraoperative core hypothermia. J Clin Anesth. 1995 Aug;7(5):359-66. doi: 10.1016/0952-8180(95)00028-g. PMID 7576669
- [Background] Frank SM, el-Gamal N, Raja SN, Wu PK. alpha-Adrenoceptor mechanisms of thermoregulation during cold challenge in humans. Clin Sci (Lond). 1996 Nov;91(5):627-31. doi: 10.1042/cs0910627. PMID 8942402
- [Background] Frank SM, Fleisher LA, Olson KF, Gorman RB, Higgins MS, Breslow MJ, Sitzmann JV, Beattie C. Multivariate determinants of early postoperative oxygen consumption in elderly patients. Effects of shivering, body temperature, and gender. Anesthesiology. 1995 Aug;83(2):241-9. doi: 10.1097/00000542-199508000-00002. PMID 7631944
- [Background] Frank SM, Higgins MS, Fleisher LA, Sitzmann JV, Raff H, Breslow MJ. Adrenergic, respiratory, and cardiovascular effects of core cooling in humans. Am J Physiol. 1997 Feb;272(2 Pt 2):R557-62. doi: 10.1152/ajpregu.1997.272.2.R557. PMID 9124478
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Du YT, Li YW, Zhao BJ, Guo XY, Feng Y, Zuo MZ, Fu C, Zhou WJ, Li HJ, Liu YF, Cheng T, Mu DL, Zeng Y, Liu PF, Li Y, An HY, Zhu SN, Li XY, Li HJ, Wu YF, Wang DX, Sessler DI; Peking University Clinical Research Program Study Group. Long-term Survival after Combined Epidural-General Anesthesia or General Anesthesia Alone: Follow-up of a Randomized Trial. Anesthesiology. 2021 Aug 1;135(2):233-245. doi: 10.1097/ALN.0000000000003835. PMID 34195784
- [Background] Mehlen P, Puisieux A. Metastasis: a question of life or death. Nat Rev Cancer. 2006 Jun;6(6):449-58. doi: 10.1038/nrc1886. PMID 16723991
- [Background] Sessler DI. Long-term consequences of anesthetic management. Anesthesiology. 2009 Jul;111(1):1-4. doi: 10.1097/ALN.0b013e3181a913e1. No abstract available. PMID 19512884
- [Background] Beilin B, Shavit Y, Razumovsky J, Wolloch Y, Zeidel A, Bessler H. Effects of mild perioperative hypothermia on cellular immune responses. Anesthesiology. 1998 Nov;89(5):1133-40. doi: 10.1097/00000542-199811000-00013. PMID 9822001
- [Background] Frank SM, Higgins MS, Breslow MJ, Fleisher LA, Gorman RB, Sitzmann JV, Raff H, Beattie C. The catecholamine, cortisol, and hemodynamic responses to mild perioperative hypothermia. A randomized clinical trial. Anesthesiology. 1995 Jan;82(1):83-93. doi: 10.1097/00000542-199501000-00012. PMID 7832339
- [Background] Yucel Y, Barlan M, Lenhardt R, Kurz A, Sessler DI. Perioperative hypothermia does not enhance the risk of cancer dissemination. Am J Surg. 2005 Jun;189(6):651-5. doi: 10.1016/j.amjsurg.2005.03.002. PMID 15910714
- [Background] Cao SJ, Zhang Y, Zhang YX, Zhao W, Pan LH, Sun XD, Jia Z, Ouyang W, Ye QS, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yu JB, Liu ZH, Yin N, Li XY, Ma JH, Li HJ, Wang MR, Sessler DI, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Delirium in older patients given propofol or sevoflurane anaesthesia for major cancer surgery: a multicentre randomised trial. Br J Anaesth. 2023 Aug;131(2):253-265. doi: 10.1016/j.bja.2023.04.024. Epub 2023 Jun 4. PMID 37474241
- [Background] Wang M, Singh A, Qureshi H, Leone A, Mascha EJ, Sessler DI. Optimal Depth for Nasopharyngeal Temperature Probe Positioning. Anesth Analg. 2016 May;122(5):1434-8. doi: 10.1213/ANE.0000000000001213. PMID 26974019
- [Background] Cipolla C, Lugo G, Tartari F, Giannini A, Monterastelli G, D'Antuono G. [Clinical, diagnostic and therapeutic aspects of non-allergic forms of rhinitis: non-allergic rhinitis with eosinophilia syndrome and vasomotor rhinitis]. Minerva Med. 1986 Feb 18;77(5-6):145-8. Italian. PMID 2936989
- [Background] Torossian A; TEMMP (Thermoregulation in Europe Monitoring and Managing Patient Temperature) Study Group. Survey on intraoperative temperature management in Europe. Eur J Anaesthesiol. 2007 Aug;24(8):668-75. doi: 10.1017/S0265021507000191. Epub 2007 Apr 11. PMID 17425815
- [Background] Matsukawa T, Sessler DI, Sessler AM, Schroeder M, Ozaki M, Kurz A, Cheng C. Heat flow and distribution during induction of general anesthesia. Anesthesiology. 1995 Mar;82(3):662-73. doi: 10.1097/00000542-199503000-00008. PMID 7879935
- [Background] Matsukawa T, Sessler DI, Christensen R, Ozaki M, Schroeder M. Heat flow and distribution during epidural anesthesia. Anesthesiology. 1995 Nov;83(5):961-7. doi: 10.1097/00000542-199511000-00008. PMID 7486181
- [Background] Wong PF, Kumar S, Bohra A, Whetter D, Leaper DJ. Randomized clinical trial of perioperative systemic warming in major elective abdominal surgery. Br J Surg. 2007 Apr;94(4):421-6. doi: 10.1002/bjs.5631. PMID 17380549
- [Background] Vanni SM, Braz JR, Modolo NS, Amorim RB, Rodrigues GR Jr. Preoperative combined with intraoperative skin-surface warming avoids hypothermia caused by general anesthesia and surgery. J Clin Anesth. 2003 Mar;15(2):119-25. doi: 10.1016/s0952-8180(02)00512-3. PMID 12719051
- [Background] Kim JY, Shinn H, Oh YJ, Hong YW, Kwak HJ, Kwak YL. The effect of skin surface warming during anesthesia preparation on preventing redistribution hypothermia in the early operative period of off-pump coronary artery bypass surgery. Eur J Cardiothorac Surg. 2006 Mar;29(3):343-7. doi: 10.1016/j.ejcts.2005.12.020. Epub 2006 Jan 24. PMID 16434206
- [Background] Just B, Trevien V, Delva E, Lienhart A. Prevention of intraoperative hypothermia by preoperative skin-surface warming. Anesthesiology. 1993 Aug;79(2):214-8. doi: 10.1097/00000542-199308000-00004. PMID 8251019
- [Background] Camus Y, Delva E, Sessler DI, Lienhart A. Pre-induction skin-surface warming minimizes intraoperative core hypothermia. J Clin Anesth. 1995 Aug;7(5):384-8. doi: 10.1016/0952-8180(95)00051-i. PMID 7576673
- [Background] Bock M, Muller J, Bach A, Bohrer H, Martin E, Motsch J. Effects of preinduction and intraoperative warming during major laparotomy. Br J Anaesth. 1998 Feb;80(2):159-63. doi: 10.1093/bja/80.2.159. PMID 9602578
- [Background] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936
- [Background] Rajek A, Greif R, Sessler DI, Baumgardner J, Laciny S, Bastanmehr H. Core cooling by central venous infusion of ice-cold (4 degrees C and 20 degrees C) fluid: isolation of core and peripheral thermal compartments. Anesthesiology. 2000 Sep;93(3):629-37. doi: 10.1097/00000542-200009000-00010. PMID 10969294
- [Background] Horn EP, Sessler DI, Standl T, Schroeder F, Bartz HJ, Beyer JC, Schulte am Esch J. Non-thermoregulatory shivering in patients recovering from isoflurane or desflurane anesthesia. Anesthesiology. 1998 Oct;89(4):878-86. doi: 10.1097/00000542-199810000-00012. PMID 9778005
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774